CLINICAL TRIAL: NCT00075179
Title: Phase IV, Open Labeled Study to Test the Effectiveness of Nesiritide in Reversing Pulmonary Hypertension in Patients Who Will be Undergoing CardioThoracic Surgery
Brief Title: Natrecor in Pulmonary Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0562
Record Dates: First submitted 2004-01-05; First posted 2004-01-06 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Hypertension; Cancer; Lung Disease; Cardiothoracic Surgery
Keywords: Pulmonary hypertension; cancer; lung cancer; lung disease; cardiothoracic surgery; Nesiritide; Natrecor; CV Surgery; Lung Tumor
MeSH Terms: conditions — Hypertension, Pulmonary; Neoplasms; Lung Diseases; Lung Neoplasms | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nesiritide (Experimental): Nesiritide 0.01 mcg/kg/min by vein over 30 minutes during right heart catheterization procedure.
  Interventions: Drug: Nesiritide (Natrecor); Procedure: Right Heart Catheterization

INTERVENTIONS:
Drug: Nesiritide (Natrecor) — Given initially as a bolus (2 mcg/kg) and than infused for 30 minutes (0.01 mcg/kg/min) during right heart catheterization.
Procedure: Right Heart Catheterization — Small tubes placed in neck vein to heart as means of measuring pressure in heart and lungs; treatment with nesiritide delivered during procedure.

SUMMARY:
The goal of this clinical research study is to learn if the drug nesiritide (Natrecor) is effective in lowering the pressure in your lungs.

The primary objective of this study is to establish that Nesiritide (Natrecor) is effective in reducing pulmonary hypertension (PHTN) acutely as measured by a 20% reduction in the mean pulmonary arterial (PA) pressure. The secondary objectives will include: improvement in pulmonary vascular resistance (PVR), patient symptoms, exercise tolerance, frequency of toxicity, and surgeon's willingness to proceed with operation.

DETAILED DESCRIPTION:
Patients with high pressure in their lungs often have many symptoms such as, shortness of breath, low energy, and fatigue. Decreasing the pressure in the lungs may help these patients feel better. The drug nesiritide was designed to help treat heart failure, however, it may also help to decrease the pressure in the lungs.

Before treatment, you will be asked questions about your medical history and about any medications you are currently taking. You will have a focused physical exam. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart). You will have an ultrasound on your heart called an echocardiogram to measure the pressures in your lungs and your ability to breathe will be evaluated. With the aid of the research nurse, you will have a 6-minute walk test if you are able. You may stop or sit down at any time during the test. This test is being done to evaluate your energy level. You will also be asked to complete a questionnaire about your symptoms. This questionnaire will take no longer than 10 minutes to complete.

In order to measure the pressure in your lungs, you will have a procedure called a "right heart catheterization". This is a procedure that may have been done as part of your standard of care if you were not enrolled in this study. For this procedure, a small tube will be placed in a vein in your neck. A longer tube will be inserted into the first tube and fed through the vein and into your heart. This tube will be used to measure the pressure in your heart and lungs. If the pressure in your lungs is above a certain level, you will receive treatment with nesiritide during the right heart catheterization procedure. Nesiritide will be given by vein over 30 minutes. After treatment, the pressure in your heart and lungs will be measured again. You will be awake during this procedure and lying flat on your back. An anesthetic will be used to numb the area of your neck where the tube is placed. The entire procedure (including treatment) should take no longer than 2 hours. When complete, the tubes will be removed.

Within 15 minutes of the end of the procedure, the 6-minute walk test (if you are able) and the questionnaire about your symptoms will be repeated and your breathing will be reassessed.

You will also have around 2 teaspoons of blood collected for special lab tests. These tests are being done to check for certain molecules in your blood. The blood that is leftover after these tests may be stored in a freezer.

Around 30 days after the procedure, you will have a follow-up visit scheduled or contacted by phone. At this visit, you will have a complete physical exam done by the doctor, and possibly have blood work done if required by the doctor as part of your routine care. There will be no additional blood work done for study purposes.

This is an investigational study. Nesiritide is FDA approved and is commercially available only for the treatment of heart failure. However, the use of nesiritide in this study is experimental. Around 20 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 85 years old.
2. Evidence of underlying lung disease by history and physical and/or chest x-ray and/or pulmonary function testing (PFT's).
3. PHTN documented by Doppler Echocardiography ( Done with in last 30 days)
4. Must be able to give an informed consent.

Exclusion Criteria:

1. Patients with clinically significant hypotension (defined as a systolic blood pressure (SBP) <90).
2. Active infection or sepsis as defined by fever and need for IV antibiotics.
3. Creatinine greater than 3.0 mg/dl
4. Significant valvular disease as a cause for the PHTN.
5. Severe Thrombocytopenia (as defined by platelets less than 20,000 or INR > 1.6.
6. Left Ventricle Ejection Fraction (LVEF) <40% (must be done with in the last 30 days prior to signing consent).
7. Hypersensitivity to nesiritide or any of it's components.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-12-31 (Actual); Primary Completion 2006-03-28 (Actual); Study Completion 2006-03-28 (Actual)

PRIMARY OUTCOMES:
Number Patients with 20% reduction in mean pulmonary arterial (PA) pressure to measure pulmonary hypertension (PHTN) | Baseline and 15 and 30 minutes after end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Lenihan, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center, Department of Cardiology — http://www.mdanderson.org/departments/cardiology/